CLINICAL TRIAL: NCT00444015
Title: Phase I Trial Evaluating the Epidermal Growth Factor Receptor Inhibitor Erlotinib in Combination With the SRC Kinase Inhibitor Dasatinib for Patients With Recurrent Non-small Cell Lung Cancer (NSCLC)
Brief Title: Phase I Dasatinib/Erlotinib in Recurrent Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14984; BMS Protocol Number: CA180080 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2011-06

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: Erlotinib; Dasatinib; Epidermal growth factor receptor (EGFR); Tyrosine kinase; NSCLC; Pharmacokinetics (PK); Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose Escalation (Experimental)
  Interventions: Drug: Erlotinib in combination with Dasatinib

INTERVENTIONS:
Drug: Erlotinib in combination with Dasatinib — 6 Cycles @ 28 Days
  Other Names: Tarceva™; SPRYCEL®

SUMMARY:
This is a single site phase I dose escalation trial of the epidermal growth factor receptor inhibitor Erlotinib with the SRC tyrosine kinase inhibitor Dasatinib in patients with previously treated advanced stage (Stage IIIB/IV disease) Non-Small Cell Lung Cancer (NSCLC). The treatment regimen consists of Erlotinib tablets starting Day 1 and Dasatinib tablets starting Day 9 for a 28-day cycle. If there are no Dose Limiting Toxicities (DLTs), dose escalation continues. The recommended phase II dose for this combined treatment will be defined and patients will be treated at the recommended phase II dose to confirm tolerability.

DETAILED DESCRIPTION:
This is a single site Phase I dose escalation trial of the epidermal growth factor receptor inhibitor Erlotinib with the SRC tyrosine kinase inhibitor Dasatinib in patients with previously treated advanced stage (Stage IIIB/IV disease) Non-Small Cell Lung Cancer (NSCLC). The screening evaluation will consist of a medical history including dates/description of your initial NSCLC diagnosis and documentation of any previous treatment. There will also be a physical examination including vital signs, height, weight, Eastern Cooperative Oncology Group (ECOG)performance status, blood draws for Complete Blood Count (CBC) and Complete Metabolic Panel (CMP) tests, neurological examination, a pregnancy test for female patients of childbearing potential, and (if applicable) any observable tumor measurements all within 14 days before study enrollment. A screening Electrocardiogram (EKG) as well as clinical testing to evaluate all known sites of malignant lesions, including Computed Tomography (CTs) of the chest and upper abdomen, the adrenal glands; ultrasound; or radionuclide scans of the bones; and/or other radiographic studies should be performed within 30 days prior to enrollment.

The treatment regimen consists of Erlotinib tablets starting Day 1 and Dasatinib tablets starting Day 9 for a 28-day cycle. If there are no DLTs, dose escalation continues. Patients continuing on therapy past two cycles will be seen by the treating physician every 4 weeks and will have complete History and Physical (H&P), CBC, and CMP. Tumor measurement and response assessment will occur every 6-8 weeks. Dasatinib and Erlotinib will be continued until progression of disease, unacceptable toxicity, or patient request.

The recommended phase II dose for this combined treatment will be defined and patients will be treated at the recommended phase II dose to confirm tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented diagnosis of NSCLC that is advanced/metastatic (Stage IIIB/IV).
* Written informed consent.
* The presence of progressive and measurable disease as defined by the -Response Evaluation Criteria in Solid Tumors (RECIST)
* Performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) Scale
* Have discontinued all previous systemic therapies for cancer, for at least 14 days prior to study entry and have had previous first line chemotherapy, have recovered from all acute effects of the therapies, and are considered for further chemotherapy, radiotherapy, or other investigational therapy after they have relapsed or progressed on previous treatment.
* Exhibit patient compliance and geographic proximity that allow for adequate follow-up.
* Adequate bone marrow reserve and organ function as follows:

  * Neutrophil count >1.5 x 10 to the 9th power/L and platelets > 100 x 10 to the 9th power/L.
  * Hepatic: total bilirubin less than or equal to 1.5 times upper limit of normal (ULN)
  * Alanine transaminase (ALT) and aspartate transaminase (AST) less than or equal to 2.5 times ULN (or less than or equal to 5 times ULN in case of known liver involvement
  * Renal: Serum Creatinine less than or equal to 1.5 times upper limit of normal (ULN)
* Reproductive potential must be either terminated (by surgery, radiation, or menopause) or attenuated by the use of an approved contraceptive method during and for 3 to 6 months following the study.
* At least 18 years of age.
* Agrees to discontinue St. Johns Wort while receiving dasatinib therapy
* Agrees that IV bisphosphonates will be withheld for the first 8 weeks of dasatinib therapy due to risk of hypocalcemia.

Exclusion Criteria:

* Prior treatment with EGFR tyrosine kinase inhibitors or EGFR targeting agent
* Have received treatment within the last 28 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Have previously completed or withdrawn from this study or any other study investigating Dasatinib.
* Pregnant or breastfeeding.
* Documented central nervous system or leptomeningeal metastasis (brain metastasis) at the time of study entry. Patients with prior brain metastasis may be considered if they have completed their treatment for brain metastasis, no longer require corticosteroids, and are asymptomatic.
* Serious concomitant disorder, including active bacterial, fungal, or viral infection, incompatible with the study (at the discretion of the investigator).
* Uncorrected electrolyte disorder, including potassium <3.0 mEq/L).
* Gastrointestinal disorder that in the opinion of the study physician may affect absorption of either erlotinib or dasatinib. This also includes the inability to swallow tablets.
* Prior major surgery or radiation therapy within 14 days of initiation of treatment
* Electrocardiogram (ECG) abnormalities indicative of cardiac disease (at the discretion of the investigator).
* Uncontrolled angina, congestive heart failure or MI within six (6) months
* Diagnosed or suspected congenital long QT syndrome
* History of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
* Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec)
* Uncontrolled hypertension.
* History of significant bleeding disorder unrelated to cancer, including:

  * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
  * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
* Patients currently taking drugs that are generally accepted to have a risk of causing Torsades de Pointes including:

  * quinidine,
  * procainamide,
  * disopyramide,
  * amiodarone,
  * sotalol,
  * ibutilide,
  * dofetilide erythromycins,
  * clarithromycin,
  * chlorpromazine,
  * haloperidol,
  * mesoridazine,
  * thioridazine,
  * pimozide,
  * cisapride,
  * bepridil,
  * droperidol,
  * methadone,
  * arsenic,
  * chloroquine,
  * domperidone,
  * halofantrine,
  * levomethadyl,
  * pentamidine,
  * sparfloxacin; and
  * lidoflazine.
* Patients with chronic obstructive pulmonary disease or pleural effusions (malignant or benign) requiring chronic oxygen therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Number of Serious Adverse Events (SAEs) Reported | 3 months per patient
  Determine the safety and tolerability of erlotinib in combination with dasatinib in patients with advanced NSCLC
Determine Maximum Tolerated Dose (MTD) | 3 months per patient
  Determine the MTD of erlotinib in combination with dasatinib and the phase II dose

SECONDARY OUTCOMES:
Pharmacokinetics (PK) | 3 months per patient
  Characterize the pharmacokinetics of the erlotinib/dasatinib combination
Changes in Serum Vascular Endothelial Growth Factor (VEGF) and Interleukin(IL)-8 Pre-treatment and Post-treatment | 3 months per patient
  Assess serum angiogenic markers as pharmacodynamic markers of treatment
Number of Participants With Complete Response (CR) and Partial Response (PR) | 3 to 6 months
  Estimate the objective response rate (CR and partial response PR). Partial Response is defined as at least a 30% decrease in the sum of longest diameter (LD) of target lesions taking as reference the baseline sum LD. Complete Response is defined as disappearance of all target lesions.
Number of Participants With Progression Free Survival (PFS) | 6 months
  Estimate the 6-month progression free survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Eric B. Haura, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffiitt Cancer Center Clinical Trials Website — http://www.moffitt.org